CLINICAL TRIAL: NCT04919642
Title: A Phase II, Open Label, Multicenter Study to Evaluate the Efficacy and Safety of TT-00420 (Tinengotinib) Tablet in Adult Patients With Advanced Cholangiocarcinoma
Brief Title: Study to Evaluate the Efficacy and Safety of TT-00420 (Tinengotinib) in Cholangiocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TransThera Sciences (Nanjing), Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TT420C1206
Expanded Access: NCT06370013 (Available)
Record Dates: First submitted 2021-05-27; First posted 2021-06-09 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2023-12

CONDITIONS: Cholangiocarcinoma; FGFR2 Fusion; FGFR2 Gene Mutation; FGFR1 Alteration; FGFR3 Alteration
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A1 (Experimental): FGFR2 fusions who have failed at least one previous treatment with an FGFR inhibitor
  Interventions: Drug: TT-00420
- Cohort A2 (Experimental): FGFR2 fusions who have previously responded on at least one previous treatment with an FGFR inhibitor and discontinued due to disease progression
  Interventions: Drug: TT-00420
- Cohort B (Experimental): Other FGFR alterations, including FGFR2 mutations and FGFR1/3 alterations, including fusions
  Interventions: Drug: TT-00420
- Cohort C (Experimental): Negative for FGFR alterations (FGFR wild-type)
  Interventions: Drug: TT-00420

INTERVENTIONS:
Drug: TT-00420 — TT-00420 tablet, administered orally once daily

SUMMARY:
This study is an open-label, multicenter study to evaluate the efficacy and safety of TT-00420 tablet in adult patients with advanced cholangiocarcinoma.

DETAILED DESCRIPTION:
This is a Phase II, open-label study to evaluate the efficacy and safety of TT00420 in patients with advanced/metastatic and surgically unresectable cholangiocarcinoma (CCA) with 1) FGFR 2 fusions who failed prior FGFR inhibitor treatment, 2) FGFR2 fusions who responded on prior FGFR inhibitor treatment, 3) with other FGFR alterations, or 4) whose tumors do not contain a detectable FGFR alteration.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age, at the time of signing informed consent
2. Histologically or cytologically documented advanced/metastatic or surgically unresectable cholangiocarcinoma who have received at least one line of prior systemic chemotherapy. Patients will be assigned to 1 of 4 cohorts:

   * Cohort A1: FGFR2 fusions who have failed at least one previous treatment with an FGFR inhibitor
   * Cohort A2: FGFR2 fusions who have previously responded on at least one previous treatment with an FGFR inhibitor
   * Cohort B: other FGFR alterations, including FGFR2 mutations and FGFR1/3 alterations, including fusions
   * Cohort C: negative for FGFR alterations (FGFR wild-type)
3. At least one measurable lesion as defined by RECIST V1.1 criteria for solid tumors5
4. Documentation of FGFR gene alteration status
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Adequate organ function confirmed at screening and within 10 days of initiating treatment, as evidenced by:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
   * Hemoglobin (Hgb) ≥ 8 g/dl
   * Platelets (plt) ≥ 75 x 10^9/L
   * aspartate aminotransferase/serum glutamate oxaloacetate transaminase (AST/SGOT) and alanine aminotransferase/serum glutamate pyruvate transaminase (ALT/SGPT) ≤ 2.5 x Upper Limit of Normal (ULN) or ≤ 5.0 x ULN if liver metastases are present
   * Total bilirubin ≤ 1.5 x ULN
   * Calculated creatine clearance ≥ 50 mL/min (Cockcroft Gault formula
7. Negative pregnancy test within 72 hours before starting study treatment in all premenopausal women and women < 12 months after the onset of menopause
8. Must agree to take sufficient contraceptive methods to avoid pregnancy (including male and female participants) during the study and until at least 6 months after ceasing study treatment
9. Able to sign informed consent and comply with the protocol

Exclusion Criteria:

1. Women who are pregnant or lactating
2. Women of child-bearing potential (WOCBP) who do not use adequate birth control
3. Patients with untreated brain or central nervous system (CNS) metastases or brain/CNS metastases that have progressed (e.g. evidence of new or enlarging brain metastasis or new neurological symptoms attributable to brain/CNS metastases) Note: Patients with treated brain metastases that are off corticosteroids and have been clinically stable for 28 days are eligible for enrollment.
4. Patients with a known concurrent malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, carcinoma in situ of the cervix or other noninvasive or indolent malignancy that has previously undergone potentially curative therapy.
5. Patients with the following mood disorders as judged by the Investigator or a psychiatrist:

   * Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia; a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others)
   * ≥ CTCAE grade 3 anxiety
6. Impaired cardiac function or significant diseases, including but not limited to any of the following:

   * left ventricular ejection fraction (LVEF) < 45% as determined by multigated acquisition (MUGA) scan or echocardiogram (ECHO)
   * Congenital long QT syndrome
   * QTcF ≥ 480 msec on screening ECG
   * Unstable angina pectoris ≤ 3 months prior to starting study drug
   * Acute myocardial infarction ≤ 3 months prior to starting study drug
7. Patients with uncontrolled hypertension (defined as blood pressure of ≥ 150 mmHg systolic and/or ≥ 90 mmHg diastolic at Screening)
8. Patients with:

   * unresolved diarrhea ≥ CTCAE grade 2, or
   * impairment of gastrointestinal (GI) function, or
   * GI disease that may significantly alter the absorption of TT-00420.
9. Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g. uncontrolled hypertriglyceridemia [triglycerides > 500 mg/dL], or active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol
10. Patients who have received chemotherapy, targeted therapy, or immunotherapy ≤ 5 half-lives or 3 weeks, whichever is shorter, (6 weeks for nitrosourea or mitomycin-C) prior to starting study drug
11. Patients who have received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered from adverse events of prior therapy
12. Patients who have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from adverse events of prior therapy
13. Patients who are currently receiving treatment with therapeutic doses of warfarin sodium (Coumadin®) or any other coumarin-derivative anticoagulants
14. Patients who are currently receiving treatment with strong CYP3A inhibitors or inducers, or sensitive substrates of CYP3A4 ≤ 2 weeks prior to starting study drug.
15. Patients who are using a proton pump inhibitor within 4 days prior to the start of study therapy or a histamine-2 blocker within 2 days prior to the start of study therapy.
16. Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory; patients with well controlled HIV might be enrolled per investigator's discretion and Sponsor approval)
17. Evidence of active infection with Hepatitis B or Hepatitis C that is not adequately controlled. For patients with known prior history of Hepatitis B or Hepatitis C, enrollment may be allowed per investigator's discretion and Sponsor approval.
18. Inability to swallow or tolerate oral medication
19. Has a history or current evidence of any condition, therapy, or laboratory abnormality that, in the opinion of the investigator, might confound the results of the trial, interfere with the patient's safe participation and compliance in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) in patients with FGFR2 fusions who have failed at least one previous treatment with an FGFR inhibitor (Cohort A1) | Through study completion, an average of 9 months.
  The proportion of subjects who achieved a complete response (CR) or a partial response (PR) based on RECIST version 1.1.
ORR in patients with FGFR2 fusions who have responded (CR or PR) on at least one previous treatment with an FGFR inhibitor and discontinued due to progressive disease (Cohort A2) | Through study completion, an average of 9 months.
ORR in patients with FGFR alterations other than FGFR2 fusions (Cohort B) | Through study completion, an average of 9 months.
ORR in patients without FGFR alterations (wild-type FGFR mutation status) (Cohort C) | Through study completion, an average of 9 months.

SECONDARY OUTCOMES:
ORR in all patients with FGFR alterations (Cohorts A and B) | Through study completion, an average of 9 months.
Progression Free Survival (PFS) (All Cohorts) | From first study drug administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
Disease Control Rate (DCR) (All Cohorts) | Through study completion, an average of 9 months.
  Defined as CR + PR + stable disease (SD)
Overall Survival (OS) (All Cohorts) | From first study drug administration until the date of death from any cause, assessed up to 24 months
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment (All Cohorts) | Up to 30 days from study discontinuation
  As assessed per CTCAE version 5.0
Concentration of TT-00420 at Protocol-Specified Timepoints (All Cohorts) | From Cycle 1 to Cycle 4, an average of 4 months (each cycle is 28 days)

OTHER OUTCOMES:
Genetic Alteration Status | Through study completion, an average of 9 months
  Evaluation of biomarkers, including but not limited to, FGFR mutation status

CONTACTS AND LOCATIONS:
Overall Officials: Milind Javle, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (32):
- United States (32):
  - Providence Cancer Center, Anchorage, Alaska
  - City of Hope, Duarte, California
  - University of California, Los Angeles, School of Medicine, Santa Monica, California
  - USO Oncology Network- Rocky Mountain Cancer Centers, Denver, Colorado
  - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Chicago Medical Center - Duchossis Center for Advanced Medicine, Chicago, Illinois
  - University of Maryland - Marlene and Stewart Greenebaum Cancer Center, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Health Center, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Comprehensive Cancer Center of Nevada, Las Vegas, Nevada
  - Summit Medical Group - Florham Park Campus, Florham Park, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Ruttenberg Treatment Center - Mount Sinai, New York, New York
  - USOR Oncology Network- New York Oncology, New York, New York
  - Stony Brook University - Long Island Cancer Center, Stony Brook, New York
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - USO Oncology Network-Northwest Cancer Specialists, P.C., Portland, Oregon
  - Medical College of South Carolina, Charleston, South Carolina
  - The University of Tennessee Medical Center, Knoxville, Tennessee
  - Sarah Cannon Research Institute at Tennessee Oncology, Nashville, Tennessee
  - Methodist Dallas Medical Center, Dallas, Texas
  - Parkland Health & Hospital System, Dallas, Texas
  - University of Texas Southwestern Harold C. Simmons Comprehensive Cancer Center, Dallas, Texas
  - Houston Methodist Hospital - Outpatient Center, Houston, Texas
  - UT MD Anderson Cancer Center, Houston, Texas
  - USO Oncology Network-Texas Oncology, Tyler, Texas
  - USO Oncology Network-Virginia Oncology Associates - Brock Cancer Center - Norfolk, Norfolk, Virginia
  - USO Oncology Network-Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Javle M, Fountzilas C, Liao CY, Pelster M, Li D, Deming D, Sahai V, Fonkoua LK, Cohn A, Mantry P, Richards D, Kingsley E, Wu F, Peng P, Hennessy K, Wang H, Sun C, Ni S, Fan J, Mahipal A. Tinengotinib for adults with advanced or metastatic cholangiocarcinoma: a multicentre, open-label, phase 2 trial. Lancet Gastroenterol Hepatol. 2026 Feb;11(2):137-149. doi: 10.1016/S2468-1253(25)00230-4. Epub 2025 Dec 2. PMID 41349554